CLINICAL TRIAL: NCT01061970
Title: Efficacy and Safety of Fispemifene in the Treatment of Hypogonadal Men With Chronic Obstructive Pulmonary Disease That Are on Oral Glucocorticoid Therapy: A 4-Week, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy and Safety of Fispemifene in the Treatment of Hypogonadal Men With Chronic Obstructive Pulmonary Disease That Are on Oral Glucocorticoid Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QuatRx Pharmaceuticals Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101-50605
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Hypogonadism; Chronic Obstructive Pulmonary Disease
Keywords: Hypogonadism; Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Hypogonadism; Pulmonary Disease, Chronic Obstructive | interventions — fispemifene

INTERVENTIONS:
Drug: Fispemifene — once daily for 4 weeks

SUMMARY:
The objective of the study is to assess and compare the preliminary efficacy, safety and tolerability of fispemifene 300 mg and placebo given once daily for 4 weeks in the treatment of hypogonadal men with chronic obstructive pulmonary disease (COPD) that are on oral glucocorticoid therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has signed a written informed consent to participate in the study and has agreed to follow dosing instructions and complete all required study visits.
2. The subject has COPD as defined by post-bronchodilator FEV1/FVC <0.7 as measured at screening.
3. The subject is on a stable dose of oral glucocorticoids (dose has not changed in the past 3 months and is not anticipated to change during the subject's participation in the study)
4. The subject is a male ≥20 years of age at the time of randomization.
5. The subject has a screening total testosterone level and a confirmatory baseline total testosterone level ≤ 350 ng/dl. Testosterone levels should be determined from early morning (0700h to 0900h) specimens.
6. The subject has a serum LH level of 1.7-15.0 IU/L and an FSH level of 1.5-15.0 IU/L at the screening visit.

Exclusion Criteria:

1. Subject has elevated prolactin. (≥21.5 ng/mL or above upper limit of reference lab range)
2. Subject has evidence of Benign Prostatic Hypertrophy (BPH) with obstructive symptoms as indicated by an International Prostate Symptom Score (IPSS) of ≥15.
3. Subject has a history of or current breast cancer, prostate cancer, abnormal DRE (with suspicion of malignancy) or elevated PSA (>4 ng/ml ) or any other malignancy. History of basal cell carcinoma is allowed.
4. Subject has a clinically significant endocrine or metabolic disease (e.g. thyroid disease, type I diabetes, severe hyperlipidemia). Severe hyperlipidemia is defined as total cholesterol >300 mg/dL or triglycerides >400 mg/dL. Type II diabetes is allowed only when HbAlc level is less than 8%.
5. Subject has clinically significant cardiovascular disease, or abnormal findings on the baseline ECG, other than those related to COPD.
6. Subject has systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥85 mmHg.
7. Subject has significant polycythemia. (Hemoglobin >17.5 gm/dL or above upper limit of reference lab range)
8. Subject has current or history of severe renal or hepatic impairment.
9. Subject has current or history of thromboembolic or blood coagulation disorder.
10. Subject has current or history of cerebrovascular incident (e.g. bleeding, stroke or transient ischemic attack).
11. Subject has clinically relevant abnormal findings in any safety laboratory tests including liver enzymes (ALT, AST) more than 1.5 times the upper limit of normal for the testing laboratory or creatinine >1.4 mg/dl .
12. Subject is heterozygous or homozygous for Factor V Leiden.
13. Subject has clinically significant abnormal findings at physical examination other than those related to COPD.
14. Subject has used transdermal testosterone therapy within 14 days or intramuscular testosterone therapy within 30 days prior to screening blood draw.
15. Subject has used any form of hormone therapy affecting estrogen and/or androgen metabolism within 30 days prior to screening blood draw.
16. Subject has used any other injectable hormonal therapy (e.g. luteinizing hormone releasing hormone (LHRH)-antagonist or- agonist, growth hormone (GH) therapy) within 30 days prior to screening blood draw.
17. Subject has used any other medication affecting the Hypothalamic-Pituitary-Gonadal (HPG)-axis within 30 days prior to screening blood draw.
18. Subject has used any dietary supplements and/or herbal therapies affecting estrogen and/or testosterone metabolism or the HPG axis within 30 days prior to screening blood draw.
19. Subject is using potent inhibitors of CYP3A4 (e.g. ketoconazole, ritonavir, etc) on Day 1 or intends to use these medications during the study.
20. Subject is using potent inducers of CYP3A4 on Randomization Day 1or intends to use these medications during the study.
21. Subject is using medication metabolized by CYP2B6, CYP2C9, CYP2C19 and CYP3A4 and having a narrow therapeutic index on Day 1 or intends to use these medications during the study
22. Subject consumes more than 14 drinks containing alcohol per week. (One drink = 1.5 oz. of distilled spirits, or 12 oz. of beer, or 5 oz. of wine.).
23. Subject has a history of or current drug abuse within 6 months prior to screening visit.
24. Subject currently has untreated sleep apnea.
25. Subject has been a participant in another clinical intervention study within 30 days prior to the planned randomization on Day 1.
26. Subject has any physical or mental condition, which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
27. Subject has previously participated in this study or any other clinical study of fispemifene.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in morning total testosterone levels | from baseline to Week 4 (end of therapy)

SECONDARY OUTCOMES:
Change in total testosterone levels | from baseline to Weeks 2 and 6
Change in free testosterone, calculated free testosterone, and DHT | from baseline to Weeks 2, 4, and 6
Change in SHBG, E2, LH, FSH, and testosterone/E2 ratio | from baseline to Weeks 2, 4, and 6
Change in serum lipid levels | from screening to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Janne Komi, MD, PhD, Study Director — Hormos Medical

REFERENCES:
- [Background] Pauwels RA, Buist AS, Calverley PM, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001 Apr;163(5):1256-76. doi: 10.1164/ajrccm.163.5.2101039. No abstract available. PMID 11316667
- [Background] Wouters EF, Creutzberg EC, Schols AM. Systemic effects in COPD. Chest. 2002 May;121(5 Suppl):127S-130S. doi: 10.1378/chest.121.5_suppl.127s. PMID 12010840
- [Background] Debigare R, Marquis K, Cote CH, Tremblay RR, Michaud A, LeBlanc P, Maltais F. Catabolic/anabolic balance and muscle wasting in patients with COPD. Chest. 2003 Jul;124(1):83-9. doi: 10.1378/chest.124.1.83. PMID 12853506
- [Background] Van Vliet M, Spruit MA, Verleden G, Kasran A, Van Herck E, Pitta F, Bouillon R, Decramer M. Hypogonadism, quadriceps weakness, and exercise intolerance in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Nov 1;172(9):1105-11. doi: 10.1164/rccm.200501-114OC. Epub 2005 Aug 11. PMID 16100014
- [Background] Kamischke A, Kemper DE, Castel MA, Luthke M, Rolf C, Behre HM, Magnussen H, Nieschlag E. Testosterone levels in men with chronic obstructive pulmonary disease with or without glucocorticoid therapy. Eur Respir J. 1998 Jan;11(1):41-5. doi: 10.1183/09031936.98.11010041. PMID 9543268
- [Background] Casaburi R, Bhasin S, Cosentino L, Porszasz J, Somfay A, Lewis MI, Fournier M, Storer TW. Effects of testosterone and resistance training in men with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Oct 15;170(8):870-8. doi: 10.1164/rccm.200305-617OC. Epub 2004 Jul 21. PMID 15271690
- [Background] Ferreira IM, Verreschi IT, Nery LE, Goldstein RS, Zamel N, Brooks D, Jardim JR. The influence of 6 months of oral anabolic steroids on body mass and respiratory muscles in undernourished COPD patients. Chest. 1998 Jul;114(1):19-28. doi: 10.1378/chest.114.1.19. PMID 9674442
- [Background] Schols AM, Soeters PB, Mostert R, Pluymers RJ, Wouters EF. Physiologic effects of nutritional support and anabolic steroids in patients with chronic obstructive pulmonary disease. A placebo-controlled randomized trial. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1268-74. doi: 10.1164/ajrccm.152.4.7551381.
- [Background] Yeh SS, DeGuzman B, Kramer T; M012 Study Group. Reversal of COPD-associated weight loss using the anabolic agent oxandrolone. Chest. 2002 Aug;122(2):421-8. doi: 10.1378/chest.122.2.421. PMID 12171812
- [Background] Svartberg J, Aasebo U, Hjalmarsen A, Sundsfjord J, Jorde R. Testosterone treatment improves body composition and sexual function in men with COPD, in a 6-month randomized controlled trial. Respir Med. 2004 Sep;98(9):906-13. doi: 10.1016/j.rmed.2004.02.015. PMID 15338805